CLINICAL TRIAL: NCT03607201
Title: Comparing Clinical Profile and Outcomes of Acute Coronary Syndrome in Diabetic and Non-Diabetic Patients
Brief Title: Acute Coronary Syndrome in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Tarumanagara University (Other)
Collaborators: Cengkareng General Hospital (Other)
Responsible Party: Principal Investigator, Anthony Paulo Sunjaya, Principal Investigator, Tarumanagara University
Other Study IDs: APS006
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Acute Coronary Syndrome; Diabetes Mellitus; Heart Failure; Acute Pulmonary Edema; Cardiac Arrythmias
Keywords: acute coronary syndrome; diabetes; heart failure; acute pulmonary edema; malignant arrhythmia
MeSH Terms: conditions — Acute Coronary Syndrome; Diabetes Mellitus; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic: History of diabetes prior to Acute Coronary Syndrome
  Interventions: Other: No intervention
- Non-diabetic: No documented history of diabetes prior to Acute Coronary Syndrome
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Routine care

SUMMARY:
This study aims to compare the clinical profile and outcomes of acute coronary syndrome patients with diabetes and without diabetes.

DETAILED DESCRIPTION:
Adult patients (≥ 18 years of age) with acute coronary syndrome which are diagnosed under International Classification of Disease (ICD-10) coding of I24.9 were included in this study. The inclusion criteria are patients with primary diagnosis of I24.9 and with a complete record of prior medical and treatment history, electrocardiographic findings, cardiac marker results and outcomes. Participants were grouped into 2 groups - diabetic and non-diabetic based on history of diabetes prior to ACS. Diagnosis of ACS was made based on clinical, electrocardiographic and cardiac marker findings found in the medical record.

Data such as age, sex, ethnic, education, prior medical and treatment history, electrocardiographic and cardiac enzyme results as well as outcomes were collected from the patients' medical records. Outcomes of interest were defined as either concomitant heart failure, acute lung edema, malignant arrhythmia, mortality or combinations of them as diagnosed in the medical records. Heart failure is defined based on echocardiographic findings from the medical records. Acute Lung Edema is defined based on medical records or reported clinical findings of lung edema - rhonchi reported in 1/3 of the lungs with oxygen saturation <90%. Whereas malignant arrhythmia is defined as the presence of ventricular tachycardia (VT) or ventricular fibrillation (VF).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute Coronary Syndrome
* Presence of detail on diabetes history

Exclusion Criteria:

* Unavailability of electrocardiographic findings, cardiac marker results
* Incomplete records of prior medical and treatment history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) with acute coronary syndrome which are diagnosed under ICD-10 coding of I24.9.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Heart Failure | Through study completion, an average of 1 year
  Based on echocardiographic findings from the medical records
Malignant Arrhythmia | Through study completion, an average of 1 year
  Presence of ventricular tachycardia (VT) or ventricular fibrillation (VF)
Acute Lung Edema | Through study completion, an average of 1 year
  Based on medical records or reported clinical findings of lung edema - rhonchi reported in 1/3 of the lungs with oxygen saturation <90%.
Cardiogenic Shock | Through study completion, an average of 1 year
  Clinical Diagnosis of Cardiogenic Shock reported in medical records
Recurrent Myocardial Infarction | Through study completion, an average of 1 year
  Clinical Diagnosis of Recurrent Myocardial Infarction reported in medical records
Mortality | Through study completion, an average of 1 year
  Patient death reported in medical records

OTHER OUTCOMES:
GRACE Score | Through study completion, an average of 1 year
  GRACE (Global Registry of Acute Coronary Events) mortality risk score
TIMI Score | Through study completion, an average of 1 year
  Thrombolysis In Myocardial Infarction (TIMI) mortality risk score

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Sunjaya, Principal Investigator — Tarumanagara University
Locations (1):
- Cengkareng General Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided